CLINICAL TRIAL: NCT00409344
Title: Phase 4 Study of Dexmedetomidine for Postoperative Sedation in Patients Undergoing Repair of Thoracoabdominal Aortic Aneurysms
Brief Title: Dexmedetomidine for Postoperative Sedation in Patients Undergoing Repair of Thoracoabdominal Aortic Aneurysms
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Surgical approach changed therefore subject enrollment not possible.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Ulrich Schmidt, MD PhD, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-P-001827; IND:74068
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Results first posted 2009-09-16 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Sedation; Respiration, Artificial; Length of Stay
Keywords: Thoracoabdominal Aortic Aneurysm; Dexmedetomidine; Mechanical ventilation
MeSH Terms: conditions — Respiratory Aspiration; Aortic Aneurysm, Thoracoabdominal | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Normal Saline
  Interventions: Other: Normal Saline
- Dexmedetomidine (Active Comparator): Dexmedetomidine is a highly specific a2 agonist with prominent central nervous system and cardiovascular effects. A postoperative sedative-hypnotic agent for intensive care patients for use up to 24 hours.
  Interventions: Drug: Dexmedetomidine; Other: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine — A continuous infusion of dexmedetomidine will be started at a dose of 0.8mcg/kg/hr. This will continue for no longer than 24 hours. Four hours post extubation the study drug wii be discontinued using a standard tapering protocol: 0.6mcg/kg/hr for 4 hours then 0.4mcg/kg/hr for 4 hours, then 0.2 mcg/kg/hr for 4 hours and then 0.1mcg/kg/hr for 4 hours and then turned off.
  Other Names: No other names have been specified
  Arms: Dexmedetomidine
Other: Normal Saline — Normal Saline will be given as the placebo and will administered at 0.8mcg/kg/hr
  Other Names: No other names have been specified

SUMMARY:
The primary objective of this study is to test the hypothesis that time on the ventilator and ICU length of stay will be shorter in TAA patients given postoperative sedation with dexmedetomidine compared to those given standard sedation. Secondary endpoints are: requirement for sedatives vasoactive drugs incidence of postoperative delirium and cost analysis.

DETAILED DESCRIPTION:
Repair of thoraco-abdominal aortic aneurysms (TAA) is mostly performed in specialized centers. These centers report an operative mortality around 10%. In an analysis of 337 consecutive TAA, Cambria et al reported pulmonary (44%), cardiac, (13.8 %) renal (13.5%) and postoperative spinal cord deficit as prominent complications. Due to the extent of the surgery and the high risk of complications, all these patients require post- operative care in the Intensive Care Unit (ICU). In 2003, the operation was performed in approximately 40 patients at the Massachusetts General Hospital (MGH). The median length of stay in the ICU was 7 days (range 2-55) All patients required postoperative mechanical ventilation for greater than 48 h. During this period, a continuous intravenous infusion of propofol is normally used for sedation. Pain relief is provided by a continuous intravenous infusion of hydromorphone. This combination of sedation and analgesia is widely used at MGH and other institutions. Although very effective, it may cause respiratory depression and a deep sedative state, which may result in a prolonged requirement for mechanical ventilation. Lighter or more controllable sedation appears to be beneficial in this regard: daily wake up of intubated and sedated ICU patients decreases days on the ventilator and length of stay in the ICU.

Dexmedetomidine is a highly specific α2 agonist with prominent central nervous system (CNS) and cardiovascular effects It is FDA-approved as a postoperative sedative-hypnotic agent for intensive care patients for use up to 24 hours. The drug has hypnotic, sedative, analgesic and anxiolytic actions, and it tends to cause a mild decrease in blood pressure and heart rate. Patients or healthy volunteers sedated with dexmedetomidine alone are easily arousable and have no apparent respiratory depression. Dexmedetomidine has synergistic hypnotic and analgesic interactions with virtually all CNS depressants tested. It significantly decreases sedative and opioid requirements during and after major surgical procedures.Other potentially beneficial effects that are not as well-documented include bronchodilation and the ability to induce a more 'physiologic' sleep than other hypnotics commonly used in the ICU. Dexmedetomidine sedation may also be associated with a lower incidence of delirium.

Patients recovering from TAA surgery routinely require substantial ICU resources. If dexmedetomidine decreases the opioid and sedative requirement in these patients, it may potentially decrease the average number of days spent on the ventilator and in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* All Patients over age 18 undergoing non-emergent repair of type I-III TAA

Exclusion Criteria:

* Pregnancy
* Patients with hepatic impairment (increase of ALT or AST three times normal)
* Patient taking clonidine or tricyclic antidepressants.
* Patients taking opioids or benzodiazepines chronically (> 2 doses a day for > 1 month)
* Patients with second or third degree heart block without a pacer
* Patients undergoing emergency repair of TAA
* Intraoperative cardiac arrest
* Intraoperative massive blood loss (>10 l)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schmidt, MD,PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period 10/10/2006 to 1/1/2008 from a surgical intensive care unit in a tertiary hospital.
Pre-assignment Details: Unable to enroll participants due to hepatic impairment and many patients taking tricyclic antidepressants.
Groups:
- Saline: This group will recive saline
- Dexmedetomidine: This group will receive dexmedetomidine
Period: Overall Study
Arm/Group | Saline | Dexmedetomidine
Started | 0 (No participants enrolled) | 0 (No participants enrolled)
Completed | 0 (No participants were enrolled to completion) | 0 (No participants were enrolled to completion)
Not Completed | 0 | 0
Not completed — no enrollment | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline | Dexmedetomidine | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to a Successful Spontaneous Breathing Trial.
Description: Did not achieve this primary outcome due to no enrollment of participants. Unable to measure this outcome.
Time Frame: 1/1/2008
Measure: Number; unit: hours
Arm/Group | Saline | Dexmedetomidine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Secondary Endpoints Include:Amount of Sedative and Opiates Given
Description: Did not achieve this outcome due to no enrollment of participants
Time Frame: 1/1/2008
Measure: Number; unit: milligram of sedative an opiate
Arm/Group | Saline | Dexmedetomidine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Extubation
Description: Did not achieve this outcome due to no enrollment of participants
Time Frame: 1/1/2008
Measure: Number; unit: hours
Arm/Group | Saline | Dexmedetomidine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Amount of Vasoactive Substances Used to Achieve Hemodynamic Stability
Description: Did not achieve this outcome due to no enrollment of participants, unable to measure this outcome
Time Frame: 1/1/2008
Measure: Number; unit: participants
Arm/Group | Saline | Dexmedetomidine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Pharmaco-economics
Description: Did not achieve this outcome due to no enrollment of participants
Time Frame: 1/1/2008
Measure: Number; unit: participants
Arm/Group | Saline | Dexmedetomidine
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Incidence of Delirium; Number of Shifts During Which Delirium Was Diagnosed
Description: Did not achieve this outcome due to no enrollment of participants. Was unable to measure this outcome.
Time Frame: 1/1/2008
Measure: Number; unit: participants
Arm/Group | Saline | Dexmedetomidine
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Intensive Care Unit Length of Stay
Description: The number of days each patient was in the Intensive Care Unit. Unable to measure this outcome due to no enrollment of participnats.
Time Frame: 1/1/2008
Measure: Number; unit: Days
Arm/Group | Saline | Dexmedetomidine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Saline | Dexmedetomidine

LIMITATIONS AND CAVEATS:
Unable to enroll participants into the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes